CLINICAL TRIAL: NCT01414413
Title: Home Assessment and Initiation of ART: a Cluster-randomised Trial in Blantyre, Malawi
Brief Title: Home Assessment and Initiation of Antiretroviral Therapy for HIV in Malawi
Acronym: CONDA-YAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kamuzu University of Health Sciences (Other); London School of Hygiene and Tropical Medicine (Other); Ministry of Health and Population, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MLW-089673; WT089673/B/09/Z (Other Grant/Funding Number: Wellcome Trust, UK)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: HIV
Keywords: HIV; AIDS; Antiretroviral therapy; Community-based study; Cluster-randomised trial; HIV testing; Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home assessment and initiation of ART (Experimental): Participants with a positive home-based HIV test result will receive a home visit from a study nurse who will complete the following on the first home visit:
  * Confirmatory fingerprick HIV testing
  * TB symptom screening
  * ART eligibility assessment (Word Health Organization clinical staging, sampling of blood for measurement of CD4 count and treatment education)
  At a second home visit (within 5 days), participants who are ART eligible (as defined in National ART guidelines) will be initiated onto ART (using National Treatment Programme ART regimens).
  Following home initiation of ART, participants in the intervention arm will receive detailed counselling from the study nurse about the need to attend their first 2-week follow-up appointment at the primary health care clinic that serves their household's residence. They will receive a referral slip detailing the date, time and place of their appointment.
  Interventions: Other: Home assessment and initiation of ART
- Clinic-based ART assessment and initiation (Other): Participants who meet eligibility criteria and reside in a cluster that has been allocated to the control arm of this study will receive supported access to ART care through the primary care system for confirmation of HIV status and entry into HIV following disclosure to the resident community counsellor. HIV care, including ART, will be started from the primary care clinic.
  Interventions: Other: Clinic-based ART assessment and initiation

INTERVENTIONS:
Other: Home assessment and initiation of ART — Home-based ART eligibility assessment (WHO staging, CD4 count measurement and educational treatment preparation) and initiation.
  Arms: Home assessment and initiation of ART
Other: Clinic-based ART assessment and initiation — Participants who meet eligibility criteria and reside in a cluster that has been allocated to the control arm of this study will receive supported access to ART care through the primary care system for confirmation of HIV status and entry into HIV following disclosure to the resident community counsellor.
  Arms: Clinic-based ART assessment and initiation

SUMMARY:
Despite increasing availability of antiretroviral therapy (ART) for HIV in high prevalence countries, the majority of people with HIV infection still initiate treatment at an advanced stage of disease. This leads to a high risk of death soon after HIV diagnosis. Prompt HIV diagnosis is, therefore, necessary for both individual and public health benefit and is being strongly promoted as international and national policy in Malawi. However timely HIV diagnosis may not in itself be sufficient to ensure ART initiation: this is reflected by the relatively high proportion of individuals who defer treatment-seeking for months or years following diagnosis of HIV.

Here the researchers investigate the extent to which home assessment and initiation of ART adds to the effectiveness of a home-based HIV testing and counseling strategy, using entry to, adherence with, and retention in HIV care as the outcome of interest.

ELIGIBILITY:
Inclusion Criteria:

* Usual resident of an eligible cluster
* Has had a positive HIV test (regardless of source) and requests facilitated access to HIV care from the resident community counsellor
* Confirmatory HIV test is positive
* No previous ART treatment, or less than one month's treatment in the past (including PMTCT interventions) and not currently receiving HIV care
* No contraindications to receiving ART (as defined by Integrated Management of Adult Illnesses, HIV Department, WHO)
* No acute danger signs requiring hospital referral
* Aged 18 years or older
* Written or witnessed informed consent to participate in the study

Exclusion Criteria:

* Not a usual resident of an eligible cluster
* No previous HIV test, or HIV infection not confirmed by home-based ART nurse
* Already receiving ART, or has had more than 1 month's treatment in the past
* Known contraindication to firstline ART (known hypersensitivity, renal failure, chronic liver disease)
* Acute danger sign present (as defined by Integrated Management of Adult Illnesses, HIV Department, WHO)
* Age younger than 18 years
* Not willing to accept home-based ART initiation
* Suspected or confirmed TB disease will not be an exclusion criteria, but will be an indication for deferral, until completion of the screening algorithm, with initiation of TB treatment if indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16660 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter MacPherson, MBChCB MPH, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Malawi-Liverpool-Wellcome Trust Clinical Research Programme, Blantyre, Chichiri, Malawi

REFERENCES:
- [Derived] MacPherson P, Lalloo DG, Webb EL, Maheswaran H, Choko AT, Makombe SD, Butterworth AE, van Oosterhout JJ, Desmond N, Thindwa D, Squire SB, Hayes RJ, Corbett EL. Effect of optional home initiation of HIV care following HIV self-testing on antiretroviral therapy initiation among adults in Malawi: a randomized clinical trial. JAMA. 2014 Jul 23-30;312(4):372-9. doi: 10.1001/jama.2014.6493. PMID 25038356
- See also: Liverpool School of Tropical Medicine — http://www.lstmliverpool.ac.uk/
- See also: Wellcome Trust — http://www.wellcome.ac.uk/

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Assessment and Initiation of ART: Optional home initiation of HIV care following HIV self-testing
- Clinic-based ART Assessment and Initiation: Facility-based HIV care following HIV self-testing only
Period: Overall Study
Arm/Group | Home Assessment and Initiation of ART | Clinic-based ART Assessment and Initiation
Started | 8194 (Adult population denominator for cluster randomised trial) | 8466 (Adult population denominator for cluster randomised trial)
Completed | 8194 (Adult population denominator for cluster randomised trial) | 8466 (Adult population denominator for cluster randomised trial)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 14 clusters included in the study had a combined adult population of 16660, with 8194 adults resident in 3213 households in the OHC arm and 8466 adults resident in 3397 households in the FCO arm. Socio-demographic characteristics assessed in the baseline enumeration were well balanced between intervention groups.
Groups:
- Home Assessment and Initiation of ART: 8194 adults resident in 3213 households
- Clinic-based ART Assessment and Initiation: 8466 adults resident in 3397 households
- Total: Total of all reporting groups
Arm/Group | Home Assessment and Initiation of ART | Clinic-based ART Assessment and Initiation | Total
Number analyzed (Participants) | 8194 | 8466 | 16660
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (11.8) | 30.2 (11.4) | 30.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3942 | 4067 | 8009
  Male | 4252 | 4399 | 8651

OUTCOME MEASURES:

1. Primary Outcome: ART Initiation
Description: Comparison between study arms of the proportion of all resident adults (per capita, and irrespective of HIV status or participation in home-based HIV testing intervention) who initiate ART during the first 6 months of the home-based HIV-testing intervention.
Time Frame: First six months following introduction of home-based HIV testing
Measure: Number; unit: participants
Arm/Group | Home Assessment and Initiation of ART | Clinic-based ART Assessment and Initiation
Number analyzed (Participants) | 8194 | 8466
participants | 181 | 63

2. Secondary Outcome: Uptake of Home-based HIV Testing
Description: Comparison between study arms of the proportion of all resident adults who request HIV testing (either as standard HTC or as supervised HIV self-testing) from the resident community counsellor during the first year of the study.
Time Frame: The first 6-months following home assessment and initiation of ART being made available
Measure: Number; unit: participants
Arm/Group | Home Assessment and Initiation of ART | Clinic-based ART Assessment and Initiation
Number analyzed (Participants) | 8194 | 8466
participants | 5287 | 4433

3. Secondary Outcome: Reporting of HIV-positive Results
Description: Comparison of the proportion of all cluster adults confiding HIV-positive results to the resident community counsellor between study arms during the 1-year study period
Time Frame: The first 6-months following availability of home-based HIV testing
Measure: Number; unit: participants
Arm/Group | Home Assessment and Initiation of ART | Clinic-based ART Assessment and Initiation
Number analyzed (Participants) | 8194 | 8466
participants | 490 | 278

4. Secondary Outcome: Loss to Retention
Description: Comparison between study arms of the proportion of participants who initiate ART during the first 6-months of the HIV-testing intervention who are lost to retention within 6 months after initiating ART 6-months
Time Frame: The first 6-months following availability of home-based HIV testing
Measure: Number; unit: participants
Arm/Group | Home Assessment and Initiation of ART | Clinic-based ART Assessment and Initiation
Number analyzed (Participants) | 181 | 63
participants | 52 | 15

5. Secondary Outcome: Adherence to ART
Description: Comparison between study arms of the proportion of HIV-positive participants who are adherent to ART during the 1-year study period
Time Frame: First 6-months following availability of home-based HIV testing
Reporting Status: Not Posted

6. Secondary Outcome: Adult Mortality
Description: Comparison between study arms of non-traumatic and HIV-related adult (15-49) mortality rates during the first 6 months of the HIV-testing intervention
Time Frame: The first 6-months following availability of home-based HIV testing
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Home Assessment and Initiation of ART | Clinic-based ART Assessment and Initiation
Serious Adverse Events (participants affected / at risk) | 0/8194 | 0/8466
Other Adverse Events (participants affected / at risk) | 0/8194 | 0/8466

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes